CLINICAL TRIAL: NCT05392010
Title: Assessment of Clinical Practice of Mechanical Ventilation After COVID-19 Pan-demic Among 57 Countries: A Systematic Analysis for the Global BurdEn of Me-chanIcal VeNtilatIon (GEMINI Study) 2022, From VENTILAGROUP.
Brief Title: Global BurdEn of MechanIcal VeNtilatIon (GEMINI). VeNtilatIon (GEMINI Study) 2022 for VENTILAGROUP.
Acronym: GEMINI
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: Spanish Research Center for Respiratory Diseases (Other)
Responsible Party: Principal Investigator, Oscar Penuelas, MD, Principal Investigator. Clinical Chief Intensive Care Unit, Hospital Universitario Getafe
Other Study IDs: GEMINI/0422
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Mechanical Ventilation; Usual Care; Noninvasive Positive Pressure Ventilation; High Flow Oxygen Therapy
Keywords: mechanical ventilation; mortality; clinical variability; precision medicine; critical illness; frailty; acute respiratory failure
MeSH Terms: conditions — Critical Illness; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ventilated critically ill patients: All consecutive adult patients (≥ 18 years old) who are admitted to the ICU and require invasive mechanical ventilation (endotracheal tube or tracheostomy) longer than 12 hours. 2. Adult patients admitted to the ICU and require advanced respiratory support (high flow oxygen nasal cannula [HFONC], or noninvasive ventilation [NIV] BIPAP or CPAP with oronasal, nasal, helmet or facial mask) with acute respiratory failure defined as PaO2/ fraction of inspired oxygen (FiO2), [PaO2/FiO2] ratio <300, or the pulse oximetric saturation (SpO2/FiO2 ) ratio < 315 for more than 1 hour.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
BACKGROUND: Changes in the clinical practice of mechanical ventilation during and after the coronavirus pandemic (COVID-19) worldwide could influence the clinical outcomes of critically ill patients with mechanical ventilation due to a generalization of these changes. Thus, the variability of the clinical response of different strategies in critically ill patients could be related to the existence of unidentified phenotypes that would be related to an increased risk of mortality and functional deterioration at the medium term.

OBJECTIVES: The main objective will be to evaluate the worldwide clinical practice of mechanical Ventilation in critically ill patients, as well as the medium-term clinical outcomes for the description of phenotypes of critically ill patients treated with mechanical ventilation.

The analysis of phenotypes and unsupervised pattern recognition over time could help to predict relevant clinical outcomes. This approach could improve personalized and precision medicine applicable to the ventilated patient. METHODOLOGY: An observational, prospective, non-interventional, international, and multicenter study will be carried out that will include adult critically ill patients requiring invasive or non-invasive mechanical ventilation for more than 12 hours. Analyzes of the variability of mortality and functional impairment at six months will be performed. Likewise, artificial intelligence analyzes ("machine learning" and "neural networks") will be carried out.

DETAILED DESCRIPTION:
Patient Population and Participating Centers Research personnel prospectively will follow up all newly admitted adult patients admitted in the ICU who received ventilator support. A region will be defined as a country or collection of countries represented by a National Coordinator. We aimed to include a total amount of ICUs with similar characteristics (approximately 1525 ICUs) from each region accordingly to the global population of the participating country. Participating centers Recruitment for participation in GEMINI study will be by open invitation, through the Steering Committee. National Coordinators will be selected, and committed to enroll local ICUs for the inclusion of patients. Participation is entirely voluntary, with no financial incentive.

Institutional review board/ Local Ethics committees approval will be obtained by the participating institutions in accordance with local ethical regulations.Currently, the study has been approved by the Ethics Committee of the Universitary Hospital of Getafe, Madrid, Spain as a coordinating center (CEIM 22/27).

Study design This will be an observational, prospective, no interventional, international and multicenter study coordinated by Hospital universitarian from Getafe, Madrid, Spain in 52 countries (see appendix for participanting regions) and will have a inclusion period of 3 months recruitment window, and then to pick any consecutive 4 week period within that window.

The recruitment framing will start October 1st 2022 until march 31th 2023. Then, a follow-up period at six months after hospital discharge.

The project will be inscribed in a Web-based resource that will provide patients, their family members, health care professionals, researchers, and the public an easy access to information regarding the protocol (clinicaltrials.gov) before the starting of the study. Study outcomes, data collection, and statistical analyses will be established a priori and submitted for publication in a peer-review International Journal before data access.

Study Population

* Inclusion Criteria In order to include participants from different regions and countries and being comparable between them, the Steering Committee will create some clinical operative definitions for the selection of the participating ICUs from each region.

This study will be conducted in Intensive Care Units ([medical ICU], coronary ICU, surgical ICU, neurocritical ICU) that meet the following criteria:

1. ICUs that have six or more beds and/or average (during prior 12 months) of more than 30% of the patients admitted requiring mechanical ventilation.
2. ICUs that have staff specialists in Intensive Care Medicine, or visiting physicians with intensive care training and/or physicians who have more than five years of intensive care experience.

   The INCLUSION CRITERIA FOR THE PATIENTS, as following:

   1. All consecutive adult patients (≥ 18 years old) who are admitted to the ICU and require invasive mechanical ventilation (endotracheal tube or tracheostomy) longer than 12 hours. 2. Adult patients admitted to the ICU and require advanced respiratory support (high flow oxygen nasal cannula, or noninvasive ventilation including BIPAP or CPAP modalities with oronasal, nasal, helmet or facial mask) with acute respiratory failure defined as PaO2/ fraction of inspired oxygen (FiO2), [PaO2/FiO2] ratio <300, or the pulse oximetric saturation (SpO2/FiO2 ) ratio < 315 for more than 1 hour.

   3. Adult patients in whom mechanical ventilation were started outside the study ICU at the same Institution and/or a different Institution, including Emergency Room, Operating Room (OR), /or were then transferred to the ICU at the participating center.

   ▪ Exclusion Criteria

   1. The following ICUs will be excluded:

a. Pediatric ICU. b. Post-Operators Anesthesia Recovery Room. 2. Patients less than 18 years old. 3. Patients admitted after elective surgery and who require mechanical ventilation for less than 12 hours (excepting patients who receive non-invasive ventilation). 4. Patients will be excluded if they were transferred to participating ICUs without a documented intubation time, or underwent a tracheotomy at prior to ICU admission. 5. Patients that were at participating ICUs for 24 hours or more, were readmitted during the study period. Study Protocol

1. Data from patients who meet the inclusion criteria and who are enrolled in the study will be collected according to the following situations, whichever occurs first:

   1. DAILY WITHIN 7 DAYS after the beginning of mechanical ventilation for recording clinical variables, and then for alternative days up to day 28.
   2. Until ICU discharge/or death after inclusion, whatever will come first for recording complications, events and clinical outcomes.
   3. FOLLOW-UP OF SIX MONTHS AFTER ICU DISCHARGE for long term outcomes, ONLY in those participants requiring invasive mechanical ventilation for at least 3 or more consecutive days.
2. If the patient is discharged from the hospital and subsequently readmitted and requires mechanical ventilation, this patient WILL NOT BE considered a new patient.
3. If the patient is transferred out of the ICU and requires ventilation during the same hospital stay WILL NOT BE considered a new patient.
4. Data will be collected using an electronic case report forms, through a secure online connection (Appendix).
5. The Investigator or Local Research Collaborator in each ICU will collect the data. It is crucially important that only the Local Research Collaborator become thoroughly familiar with the study objectives and data collection in each ICU. Otherwise, there is a risk that the normal routine in an ICU will be disrupted, and data collected will no longer reflect usual activities.
6. The National Coordinator for each country must be consulted regarding any protocol related questions.

   ▪ Outcomes The main outcome will be ICU mortality. The secondary outcomes will include: frailty at 6 months from hospital discharge (only for those participants requiring invasive mechanical ventilation for at least 3 consecutive days), 28-day mortality, hospital and 6-months mortality, length of ICU and hospital stay, duration of ventilatory support, free-hospital days and free-ventilator days, failure of noninvasive respiratory support, reintubation rate, tracheotomy rate, decision for withdrawal or withholding vital support rate, and ICU readmission rate.

   Other intermediate outcomes will be as: rate of complications and organ failure during ICU stay (barotrauma, delirium, ICU-acquired weakness, acute renal failure or need of replacement renal therapy, shock).

   Data collection Data regarding written directives, demographic data, comorbidities, frailty scale (baseline health will be assessed and disability in the month before ICU admission retrospectively at six months), daily screening, preferred modalities of ventilator support, ventilatory approach for liberation from mechanical ventilation, and practices of sedation or neuromuscular blockers pertaining to invasive mechanical ventilation and discontinuation will be collected daily during the period of ventilatory support.

   Case report forms (CRFs; appendix) will be electronically provided by the investigators using a secured internet based website. Data collection on admission will included demographic data and comorbid diseases. Clinical and laboratory data for simplified acute physiology score (SAPS) 3 will be reported as the worst values within 24 h after admission. A daily assessment of organ function in accordance with the sequential organ failure assessment (SOFA) score5 will be done.

   ▪ Statistical analyses Randomization This is a prospective, observational, and no intervention study, and therefore, randomization is not applicable.

   Sample size calculation Despite of the characteristics of this observational study (an international and multicenter observational study) with multiple objectives to evaluate, we will decide to include patients according with the calculation of the sample size for the main objective (ICU mortality).

   In this way, we estimated that 9,092 patients would need to be enrolled for the study to have 90% power to detect a rate of ICU mortality of 25% versus 28% in the previous study, at an overall two-sided alpha level of 0.05. By assuming 20% of missing cases, a final 10,910 patient will be required for the study.

   In addition to the statistical criterion, a hierarchical criterion will be added regarding the minimum number of cases included depending on the demographics of the participating countries, in order to obtain information on representative clinical practice. Then, the study should reach 500 cases per country with <10 million inhabitants , 500-1000 cases for countries with 11-25 million, 1000-1500 cases for countries with 26-50 million and more than 1200 cases for countries with more than 50 million inhabitants.

   The secondary objectives will be tested using the same sample size. Statistical Methods The investigators will used descriptive statistics to summarize binary (number and percentage, and continuous (mean and standard deviations (SD) and median and interquartile range [IQR], when appropriate) variables. The Kolmogorov-Smirnov test will be used, and histograms and quantile-quantile plots will be examined to verify if there were significant deviations from the normality assumption of continuous variables Student's t or Mann Whitney U tests will be use to compare continuous variables and chi-squared tests will be used for categorical variables.

   The investigators will express differences in clinical outcomes using the absolute difference with 95% confidence intervals with Yates continuity correction for binary outcomes and median (IQR) with bootstrapped 95% for continuous outcomes.

   P values will be adjusted for clustering of ICUs within hospitals by using a mixed-model framework and will be corrected for multiple testing using the Holmes-Bonferroni method.

   Residuals will be assessed to ensure the normality assumption. A logistic model with a logit link function will be used to identify baseline characteristics and factors that developed between ICU admission and clinical outcomes and complications related to the use of specific ventilatory strategies and comorbidities and frailty.

   Clustering will be accounted for by including a random effect for hospital. To identify factors associated with ICU mortality, the researchers will construct two different approaches: a multilevel logistic model with a logit link including patient variables (age, basal frailty, IMV duration, modified Sequential Organ Failure Assessment [SOFA] respiratory score, , and primary diagnosis; model 1); patient and site variables (screening, hospital type, hospital profit status, and adjusting IMV support, and region; model 2); and patient, site, and practitioner variables (model 3). On the other hand, we will develop different models of machine learning to identify clinical subphenotypes to predict clinical outcomes as ICU mortality, 6-months mortality, successful extubation or prolonged ventilatory support as main secondary outcomes.

   Adjusted model will have the best balance of variables based on discrimination (C statistic) and calibration (calibration slope and calibration-in-the-large) after performing internal bootstrap validation and finally an external validation as sensitivity analysis by taking 30% of the global cohort of included patients. The investigators will assume that missing variables in regression analyses (eg, SAPS 3 score at ICU admission, SOFA score) will be missing at random.

   These variables will be imputed using multiple imputation by chained equations. A 2-sided P values <.05 will indicate statistical significance.

   The least significant difference testing procedure will be used for pairwise comparisons.

   In-hospital death will be analyzed using multilevel logistic regression with three levels: hospital, and country. The results of fixed effects (measures of association) will be given as odds ratios (OR) with their 95% CIs and the 80% interval OR. Random effects (measures of variation) measures included the variance and its SE, the proportional change in variance, and the median OR (MOR).

   Data will be processed and analyzed in the department of Statistics department of the Hospital Universitario Ramón y Cajal (Madrid, Spain), in collaboration with the department of intensive care of Getafe University Hospital (Madrid, Spain). Analyses will be performed using Stata Software 16.0 (StataCorp LP, College Station, Texas). This study follows multidisciplinary guidelines for reporting machine learning predictive models in biomedical research. A number of classification models will be used, including logistic regression, neural networks, and ensemble models such as random forest and decision trees.

   Data collection methods All data used in this study will be routinely collected from the clinical parameters obtained daily during the ICU admission. These data will be collected by each participating center led by a local coordinator and saved in an online database created ad hoc according with legislation and in adherence with safety and confidential international legal requirements and will have a personal access for National Coordinators and local collaborators under a personal profile with username and password.

   This online database will be designed in the Hospital universitarian from Getafe. Finally, the principal investigator will store the completed, anonymous and irreversible database with a limited access during 20 years. Detailed instructions explaining the aim of the study, instructions for data collection, and definitions were available through a secured website for all participants before starting data collection and throughout the study period. The coordinating Centre will answer any additional queries on a per case basis during data collection. Validity checks will be made concurrent with data entry on the electronic CRF including plausibility checks within each variable and between variables. Data will be further reviewed by the coordinating centre for plausibility and availability of outcome parameter (death in the ICU), and any doubts will be clarified with the centre in question. There will not be on-site monitoring. However, National Coordinators will send queries to local collaborators to fulfill outliers and main missing data.

   For the purposes of this study, the world was divided into nine geographical regions:

   North America, South America, Western Europe, Eastern Europe, Middle East, south Asia, east and southeast Asia, Oceania, and Africa. Individual countries will be also classified into three income groups in accordance with their 2020 gross national income (GNI) per person, using thresholds defined by the World Bank Atlas method: (World Bank. GNI per capita, Atlas method (current US$). http://data.worldbank.org/indicator/NY.GNP.PCAP.

   CD (accessed April 5, 2022); GNI less than US$8700 was defined as low and lowermiddle income, $8700-$19400 was defined as upper-middle income, and greater than $19400 was defined as high income). Detailed instructions explaining the aim of the study, instructions for data collection, and definitions will be available through a secured website for all participants before starting data collection and throughout the study period. Any additional queries will be answered on a percase basis by the coordinating centre during data collection. Validity checks will be made concurrent with data entry on the electronic CRF including plausibility checks within each variable and between variables.

   Data monitoring Committee (DMC) A committee of three main investigators will ensure the rights and safety of participants involved in the study are protected. Main missing variables will be detected and will sent to the National Coordinators to be completed.

   Quality Control Extensive efforts will be made to ensure the quality of the data collected throughout the study. At each site, the study physicians, including review of the chart, will review the data from a randomly chosen 5 percent of screened patients and from all patients about whom the screeners had questions. Data from a random sample of 7 percent of cases were abstracted and entered into the database twice, with an error rate of less than 0.25 percent.

   The charts will be reevaluated until the final notes, laboratory test results, and other results will be completed. Complete data will be necessary to include participants in the final analysis, and we will accept participants with no missing data for the main variables or participants with missing data less than 10% for secondary variables.

   All local regulations must be met and the necessary documentation submitted to the Study Coordinating Center. Physicians from each participating country as lead national coordinators will be recruited.

   Site investigators will be also responsible for ensuring safety, anonymous data integrity and validity. The Steering Committee and National Coordinators will have full access to all the data in the study and had final responsibility for the decision to submit for publication.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (≥ 18 years old) who are admitted to the ICU and require invasive mechanical ventilation (endotracheal tube or tracheostomy) longer than 12 hours. 2. Adult patients admitted to the ICU and require advanced respiratory support (high flow oxygen nasal cannula [HFONC], or noninvasive ventilation [NIV] BIPAP or CPAP with oronasal, nasal, helmet or facial mask) with acute respiratory failure defined as PaO2/ fraction of inspired oxygen (FiO2), [PaO2/FiO2] ratio <300, or the pulse oximetric saturation (SpO2/FiO2 ) ratio < 315 for more than 1 hour. 3. Adult patients in whom mechanical ventilation were started outside the study ICU at the same Institution and/or a different Institution, including Emergency Room, Operating Room (OR), /or were then transferred to the ICU at the participating center

Exclusion Criteria:

* The following ICUs will be excluded:

  1. Pediatric ICU.
  2. Post-Operators Anesthesia Recovery Room. 2. Patients less than 18 years old. 3. Patients admitted after elective surgery and who require mechanical ventilation for less than 12 hours (excepting patients who receive non-invasive ventilation). 4. Patients will be excluded if they were transferred to participating ICUs without a documented intubation time, or underwent a tracheotomy at prior to ICU admission. 5. Patients that were at participating ICUs for 24 hours or more, were readmitted during the study period

Ages: 18 Years to 119 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to include participants from different regions and countries and being comparable between them, the Steering Committee will create some clinical operative definitions for the selection of the participating ICUs from each region.The study population will be adult critically ill patients with acute respiratory failure and need of ventilatory support (inv asive or noninvasive oxigenation support, including high flow oxygen therapy or noninvasive ventilation).
Sampling Method: Non-Probability Sample
Enrollment: 10900 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | From date of inclusion until the date of death from any cause during ICU stay, whichever came first, assessed up to 6 weeks
  rate of dead patients requiring mechanical ventilation during ICU stay

SECONDARY OUTCOMES:
hospital mortality. | From date of inclusion until the date of death from any cause during hospital stay, whichever came first, assessed up to 6 months
  rate of dead patients requiring mechanical ventilation during hospital stay
duration of mechanical ventilation. | from orotracheal intubation date until scheduled extubation date or 24 hours of unassisted respiratory support in tracheotomized patietns
  length of invasive ventilatory support
28-day mortality. | from initiacion from mechanical ventilation until 28-day hospital stay.
  rate of dead patients requiring mechanical ventilation until 28-day hospital stay
6 months mortality | from hospital discharge date until 6 months of follow-up in surviors from ICU stay.
  rate of dead patients requiring 3 days of mechanical ventilation after hospital discharge
6-months frailty. | from hospital discharge date until 6 months of follow-up in surviors from ICU stay, assessed by Clinical Frailty Scale (CFS, where values between 1-9 points, a higher scores mean a worse outcome)
  assessment of clinical frailty scale at 6-months after hospital discharge.
reintubation. | From date of orotracheal scheduled extubation until the date of reintubation from any cause during ICU stay, assessed up to 48 hours
  rate of failed extubated patients following 48 hours from scheduled extubation
ICU stay. | From date of inclusion (ICU admission) until the date of ICU discharge, assessed up to 6 weeks, including survivors and nonsurvivors from ICU
  length of ICU stay.
hospital stay. | From date of inclusion (ICU admission) until the date of hospital discharge, assessed up to 6 monthss including survivors and nonsurvivors from ICU
  length of hospital stay.
ICU free days. | events during ICU stay (from ICU admission to ICU discharge dates)
  It will defined the ICU-free days as 30 minus the number of days in the ICU (range, 0-30 days). For patients who survived and were in the ICU for less than 30 days, the ICU-free day's outcome measure was obtained by subtracting the length of the ICU stay from 30
ventilator-free days (VFD). | events during ICU stay (from ICU admission to ICU discharge dates) From date of orotracheal intubation until the date of unassisted positive pressure ventilation, either without orotracheal tube or tracheal cannula, assessed up to 6 months
  VFD will be defined as follows:
  * VFDs = 0 if subject dies within 28 days of mechanical ventilation.
  * VFDs = 28 - x if successfully liberated from ventilation x days after initiation.
  * VFDs = 0 if the subject is mechanically ventilated for >28 days
tracheotomy rate. | events during ICU stay (rate of performance for scheduled tracheotomy, assessed up to 6 months)
  rate of tracheotomized patients in those patients receiving invasive mechanical ventilation
decision for withdrawal or withholding vital support rate. | events during ICU admission through study completion, an average of 6 months.
  rate of those patients that will have a decision for withdrawal or withholding vital support rate during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Penuelas, P.h.D, Principal Investigator — Hospital Universitario de Getafe, Madrid, Spain
Locations (1):
- Intensive Care Unit, Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med. 2010 Oct;38(10):1947-53. doi: 10.1097/CCM.0b013e3181ef4460. PMID 20639743
- [Background] Carson SS, Cox CE, Holmes GM, Howard A, Carey TS. The changing epidemiology of mechanical ventilation: a population-based study. J Intensive Care Med. 2006 May-Jun;21(3):173-82. doi: 10.1177/0885066605282784. PMID 16672639
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Background] Wunsch H, Wagner J, Herlim M, Chong DH, Kramer AA, Halpern SD. ICU occupancy and mechanical ventilator use in the United States. Crit Care Med. 2013 Dec;41(12):2712-9. doi: 10.1097/CCM.0b013e318298a139. PMID 23963122
- [Background] Penuelas O, Muriel A, Abraira V, Frutos-Vivar F, Mancebo J, Raymondos K, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Ferguson ND, Del Carmen Marin M, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Amin P, Cakar N, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Esteban A. Inter-country variability over time in the mortality of mechanically ventilated patients. Intensive Care Med. 2020 Mar;46(3):444-453. doi: 10.1007/s00134-019-05867-9. Epub 2020 Jan 7. PMID 31912203
- [Background] Vincent JL, Sakr Y, Ranieri VM. Epidemiology and outcome of acute respiratory failure in intensive care unit patients. Crit Care Med. 2003 Apr;31(4 Suppl):S296-9. doi: 10.1097/01.CCM.0000057906.89552.8F. PMID 12682455
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Vincent JL, Marshall JC, Namendys-Silva SA, Francois B, Martin-Loeches I, Lipman J, Reinhart K, Antonelli M, Pickkers P, Njimi H, Jimenez E, Sakr Y; ICON investigators. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014 May;2(5):380-6. doi: 10.1016/S2213-2600(14)70061-X. Epub 2014 Apr 14. PMID 24740011
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Reddy K, Sinha P, O'Kane CM, Gordon AC, Calfee CS, McAuley DF. Subphenotypes in critical care: translation into clinical practice. Lancet Respir Med. 2020 Jun;8(6):631-643. doi: 10.1016/S2213-2600(20)30124-7. PMID 32526190
- [Background] Shah FA, Meyer NJ, Angus DC, Awdish R, Azoulay E, Calfee CS, Clermont G, Gordon AC, Kwizera A, Leligdowicz A, Marshall JC, Mikacenic C, Sinha P, Venkatesh B, Wong HR, Zampieri FG, Yende S. A Research Agenda for Precision Medicine in Sepsis and Acute Respiratory Distress Syndrome: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2021 Oct 15;204(8):891-901. doi: 10.1164/rccm.202108-1908ST. PMID 34652268
- [Background] Higgins AM, Neto AS, Bailey M, Barrett J, Bellomo R, Cooper DJ, Gabbe BJ, Linke N, Myles PS, Paton M, Philpot S, Shulman M, Young M, Hodgson CL; PREDICT Study Investigators. Predictors of death and new disability after critical illness: a multicentre prospective cohort study. Intensive Care Med. 2021 Jul;47(7):772-781. doi: 10.1007/s00134-021-06438-7. Epub 2021 Jun 5. PMID 34089063
- [Background] Hodgson CL, Udy AA, Bailey M, Barrett J, Bellomo R, Bucknall T, Gabbe BJ, Higgins AM, Iwashyna TJ, Hunt-Smith J, Murray LJ, Myles PS, Ponsford J, Pilcher D, Walker C, Young M, Cooper DJ. The impact of disability in survivors of critical illness. Intensive Care Med. 2017 Jul;43(7):992-1001. doi: 10.1007/s00134-017-4830-0. Epub 2017 May 22. PMID 28534110
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] COVID-ICU Group on behalf of the REVA Network and the COVID-ICU Investigators. Clinical characteristics and day-90 outcomes of 4244 critically ill adults with COVID-19: a prospective cohort study. Intensive Care Med. 2021 Jan;47(1):60-73. doi: 10.1007/s00134-020-06294-x. Epub 2020 Oct 29. PMID 33211135